CLINICAL TRIAL: NCT05678374
Title: Exploring Immunological Markers in Blood and Cerebrospinal Fluid Associated With Mental Fatigue in Euthyroidism After Graves' Disease- a Cross Sectional Study
Brief Title: Exploring Immunological Markers Associated With Mental Fatigue in Graves' Disease
Status: Recruiting | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: ImmunoGraves WP1
Record Dates: First submitted 2022-12-19; First posted 2023-01-10 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Graves Disease; Graves Ophthalmopathy; Mental Fatigue; Autoimmune Diseases; Thyroid Diseases
Keywords: Biomarkers; Cerebrospinal fluid in Graves' disease
MeSH Terms: conditions — Graves Disease; Graves Ophthalmopathy; Mental Fatigue; Autoimmune Diseases; Thyroid Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Graves' patients with mental fatigue: Women diagnosed with Graves 15 moths to 60 months ago with Mental Fatigue Scale score of more than 13 (maximum 42, cut of 10,5 for mental fatigue)
- Graves' patients without mental fatigue: Women diagnosed with Graves 15 moths to 60 months ago with Mental Fatigue Scale score of less than 8 (maximum 42, cut of 10,5 for mental fatigue)
- Thyroid healthy controls without mental fatigue: Women without current or previous thyroid disease and with Mental Fatigue Scale scores of less than 8

SUMMARY:
Mental fatigue occurs in many diseases and the reasons are mostly unknown. The investigators hypothesize that remaining mental fatigue after restored hyperthyroidism in Graves' disease is an autoimmune complication. The aim of this study is to explore immunological markers possibly associated with mental fatigue in Graves' disease, which the investigators plan to validate in another study (ImmunoGraves wp 2).

Using a cross-sectional study design, mental fatigue is scored using a questionnaire to find 60 patients with and 60 without mental fatigue 15-60 months after diagnosis of Graves disease. The patients and 60 thyroid healthy controls without mental fatigue are assessed for thyroid hormones, quality of life, anxiety and depression, self-evaluated stress, coping strategies, eye symptoms and background variables. SciLifeLab in Stockholm, the national facility for autoimmune profiling, has pre-set large arrays including 42000 human proteins. Serum and cerebrospinal fluid will be separately pooled and analysed for a subgroup of patients with or without mental fatigue and for a subgroup of the control group. Proteins that preferably bind to antibodies in sera and/or cerebrospinal fluid from Graves' patients with mental fatigue in comparison to non-mental fatigue patients, will be screened against the Human Protein Atlas and the Allen brain map to identify those proteins that are expressed in the brain. Antibodies at higher concentration in the mental fatigue pools compared to the group without mental fatigue will be selected for further analyses on an individual level in the whole cohort together with antibodies targeting g-protein coupled receptors, thyroid autoantibodies, cytokines and biomarkers indicating organic and structural nerve damage.

ELIGIBILITY:
Inclusion Criteria

* If patient: Graves' disease with positive TSH-receptor antibodies and thyroid hormones above the upper reference limit at diagnosis
* Diagnosis15 to 60 months ago. If recidive both episodes must have occurred within 15 months to 60 months.
* Thyroid hormones within normal range without anti thyroid drugs
* If control: No thyroid disease
* Patient and control without mental fatigue: Mental Fatigue Score ≤8 (cut off 10.5)
* Patient with mental fatigue: Mental Fatigue Score >13 and debut of symptoms of mental fatigue in parallel with debut of Graves' disease, without other obvious cause

Exclusion Criteria

* Person unable to follow protocol
* Multiple sclerosis, myalgic encephalomyelitis/chronic fatigue syndrome, any other neurological disease
* Traumatic brain injury with unconsciousness
* Other disease strongly associated with fatigue
* Pregnancy and breast-feeding
* On-going or recent systemic treatment with steroids
* Radioiodine therapy within the last 18 months

Ages: 18 Years to 72 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients are recruited from the both previous patients at the Endocrine outpatient Clinic at Sahlgrenska University Hospital in Gothenburg and from advertising. They are invited to a web based screening form where the ones eligible are contacted by study personal and eligibility criteria are checked again.
  Controls are recruited by the same way and by contacting a random sample from the population registration (based on Swedish social security number).
  Groups are matched for age, educational level and smoking habits.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2028-12-20 (Estimated); Study Completion 2028-12-20 (Estimated)

PRIMARY OUTCOMES:
Identifying autoantibodies targeting antigens occurring in the brain that are higher in Graves' disease complicated by mental fatigue than in Graves' disease not complicated by mental fatigue | Patients and controls will be examined at one occasion, for patients 15-60 months after diagnosis of Graves' disease.
  Each group will be analysed in arrays for antibodies targeting 42000 human proteins (ScilifeLabs, Stockholm). Proteins binding to antibodies in mental fatigue patients will be screened against the Human Protein Atlas (www.proteinatlas.org) and the Allen brain map (www.brain-map.org) and those expressed in the brain will be compared between groups.

SECONDARY OUTCOMES:
Identifying autoantibodies targeting antigens occurring in the brain that are higher in Graves' disease complicated by mental fatigue than in thyroid healthy controls without mental fatigue | Patients and controls will be examined at one occasion, for patients 15-60 months after diagnosis of Graves' disease.
  Each group will be analysed in arrays for antibodies targeting 42000 human proteins (ScilifeLabs, Stockholm). Proteins binding to antibodies in mental fatigue patients will be screened against the Human Protein Atlas (www.proteinatlas.org) and the Allen brain map (www.brain-map.org) and those expressed in the brain will be compared between groups.
Identifying autoantibodies targeting antigens occurring in the brain that are higher in Graves' disease not complicated by mental fatigue than in thyroid healthy controls without mental fatigue | Patients and controls will be examined at one occasion, for patients 15-60 months after diagnosis of Graves' disease.
  Each group will be analysed in arrays for Ab targeting 42000 human proteins (ScilifeLabs, Stockholm). Proteins binding to Ab in MF patients will be screened against the Human Protein Atlas (www.proteinatlas.org) and the Allen brain map (www.brain-map.org) and those expressed in the brain will be compared between groups.
Thyroid autoantibodies compared between Graves' disease complicated by mental fatigue, Graves' disease not complicated by mental fatigue and healthy controls | Patients and controls will be examined at one occasion, for patients 15-60 months after diagnosis of Graves' disease.
  Levels of thyroid autoantibodies will be analysed with the standard method of the laboratory at Sahlgrenska University Hospital.
Cytokines compared between Graves' disease complicated by mental fatigue, Graves' disease not complicated by mental fatigue and healthy controls | Patients and controls will be examined at one occasion, for patients 15-60 months after diagnosis of Graves' disease.
  Levels of cytokines will be analysed with the standard method of the laboratory at Sahlgrenska University Hospital.
Biomarkers indicating organic and structural nerve damage compared between Graves' disease complicated by mental fatigue, Graves' disease not complicated by mental fatigue and healthy controls | Patients and controls will be examined at one occasion, for patients 15-60 months after diagnosis of Graves' disease.
  Biomarkers will be analysed with the standard method of the laboratory at Sahlgrenska University Hospital.
Autoantibodies to other g-protein coupled receptors compared between Graves' disease complicated by mental fatigue, Graves' disease not complicated by mental fatigue and healthy controls | Patients and controls will be examined at one occasion, for patients 15-60 months after diagnosis of Graves' disease.
  Levels of autoantibodies to g-protein coupled receptors will be measured using enzyme-linked immunosorbent assays
Prevalence of endocrine ophthalmopathy in Graves' complicated by mental fatigue compared to prevalence of endocrine ophtalmopathy in Graves' not complicated by mental fatigue | Patients and controls will be examined at one occasion, for patients 15-60 months after diagnosis of Graves' disease.
  Prevalence defined as endocrine ophthalmopathy that has required assessment/and or follow up at ophthalmologist.
Self evaluated quality of life in relation to ophthalmopathy will be compared between patients with Graves' with and without mental fatigue and to healthy controls | Patients and controls will be examined at one occasion, for patients 15-60 months after diagnosis of Graves' disease.
  Evaluated by the validated questionnaire the Graves' Ophthalmopathy Quality of Life Questionnaire (GO QoL).
Self evaluated quality of life in relation to thyroid symptoms will be compared between patients with Graves' with and without mental fatigue and to healthy controls | Patients and controls will be examined at one occasion, for patients 15-60 months after diagnosis of Graves' disease.
  Evaluated by the validated questionnaire Thyroid-specific Patient-Reported Outcome short-form (ThyPro 39)
Self evaluated quality of life and well being will be compared between patients with Graves' with and without mental fatigue and to healthy controls | Patients and controls will be examined at one occasion, for patients 15-60 months after diagnosis of Graves' disease.
  Evaluated by the validated questionnaire Psychological General Well Being index (PGWB)
Self evaluated symptoms of anxiety and depression will be compared between patients with Graves' with and without mental fatigue and to healthy controls | Patients and controls will be examined at one occasion, for patients 15-60 months after diagnosis of Graves' disease.
  Evaluated by the validated questionnaire the Comprehensive Psychopathological Rating Scale (CPRS).
Self evaluated stress will be compared between patients with Graves' with and without mental fatigue and to healthy controls | Patients and controls will be examined at one occasion, for patients 15-60 months after diagnosis of Graves' disease.
  Evaluated by the validated questionnaire Perceived Stress Scale (PSS-14).
Coping strategies will be compared between patients with Graves' with and without mental fatigue and to healthy controls | Patients and controls will be examined at one occasion, for patients 15-60 months after diagnosis of Graves' disease.
  Evaluated by the validated questionnaire Brief cope.
Optimistic self-beliefs to cope with difficulties in life will be compared between patients with Graves' with and without mental fatigue and to healthy controls | Patients and controls will be examined at one occasion, for patients 15-60 months after diagnosis of Graves' disease.
  Evaluated by the validated questionnaire General self efficacy.
Personality traits will be compared between patients with Graves' with and without mental fatigue and to healthy controls | Patients and controls will be examined at one occasion, for patients 15-60 months after diagnosis of Graves' disease.
  Evaluated by the validated questionnaire NEO Five-Factor Inventory-3 (NEO-FFI-3).

CONTACTS AND LOCATIONS:
Overall Officials: Helena Filipsson, Principal Investigator — Institute of Medicine, Sahlgrenska Academy, University of Gothenburg
Locations (1):
- Department of Endocrinology, Sahlgrenska University Hospital, Gothenburg, Sweden